CLINICAL TRIAL: NCT00233896
Title: A Randomized, Placebo-Controlled, Multi-Center Study of Oral Beclomethasone Dipropionate With Ten Days of Prednisone for Treatment of Gastrointestinal Graft Vs. Host Disease
Brief Title: Randomized Study of Oral Beclomethasone Dipropionate With Ten Days of Prednisone for Treatment of Gastrointestinal GVHD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Enteron Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ENT 00-02
Record Dates: First submitted 2005-10-04; First posted 2005-10-06 (Estimated); Last update posted 2005-10-06 (Estimated); Status verified 2004-12

CONDITIONS: Graft Vs Host Disease; Gastrointestinal Graft-Versus-Host Disease
Keywords: Hematopoietic cell transplant; Acute graft-vs.-host disease; Gastrointestinal tract; Randomized trial; Topical corticosteroid; Beclomethasone dipropionate; Prednisone; Survival
MeSH Terms: conditions — Graft vs Host Disease | interventions — Beclomethasone; Pharmaceutical Preparations

INTERVENTIONS:
Drug: Oral beclomethasone dipropionate (drug)

SUMMARY:
Patients with gastrointestinal graft-vs.-host disease are randomized to oral beclomethasone dipropionate (BDP) 8 mg/day or identical placebo tablets for 50 days, along with a 10-day induction course of prednisone. At study day 10, patients whose symptoms of GVHD are under control undergo a rapid prednisone taper over 7 days, while study drug is continued to study day 50. After discontinuation of study drug at study day 50, patients are followed for 30 additional days, to study day 80. The primary endpoint is treatment failure by day 50, that is, a flare of the symptoms of GVHD that requires immunosuppressive therapy. Secondary endpoints are treatment failure by day 80, treatment-emergent adverse events, and survival at transplant day 200. The hypothesis to be tested is that a topically-active corticosteroid (beclomethasone dipropionate, BDP), taken orally, would allow rapid tapering of prednisone while maintaining control of intestinal GVHD.

DETAILED DESCRIPTION:
Patient selection. Patients who develop symptoms of GVHD are evaluated with endoscopy and mucosal biopsy. If biopsy specimens demonstrate histologic findings of GVHD and stool and mucosal biopsy cultures are negative for pathogens, patients are invited to participate. Patients are excluded if diarrhea exceeds one liter per day, or if skin or liver GVHD are present. All patients receive medications for GVHD prophylaxis; patients receiving corticosteroids within 30 days of study entry are excluded. Patients signed informed consent documents approved by Institutional Review Boards.

Formulation of BDP. Immediate release tablets and enteric-coated tablets, each contained 1 mg of BDP (orBec, DOR BioPharma, Miami FL). The dosing regimen was one immediate release and one enteric-coated tablet, taken orally four times daily (total daily dose, 8 mg BDP).

Stratification and randomization. A stratified allocation scheme is used to balance the treatment groups within study centers. Stratifying variables are HLA-matched sibling and use of cutaneous corticosteroids at baseline. Patients receive either BDP or identical placebo tablets.

Treatment plan. Therapy consists of study drugs plus 10 days of prednisone at an initial prednisone dose of 1 mg/kg/day. In patients with control of GVHD symptoms at Study Day 10, prednisone is tapered over 7 days, after which patients were maintained on physiologic replacement doses of prednisone. Patients who do not demonstrate adequate control of GVHD by Study Day 10 are considered treatment failures. Patients receive study drug for 50 days, or until they meet the treatment failure endpoint, or are withdrawn from the study. Patients who are declared treatment failures have study drug discontinued; subsequent treatment for GVHD is dictated by their physicians.

Definitions of treatment failure and efficacy end-points. Treatment failure is a worsening or recurrence of GVHD that requires additional immunosuppressive therapy. The primary efficacy endpoint is the time to treatment failure through Study Day 50. Secondary efficacy endpoints included time to treatment failure through Study Day 80 (30 days after discontinuation of study drug); the proportion who experience treatment failure by Study Days 10, 30, 50, and 80; and the overall survival rate at day-200 days post-transplant.

Evaluation of drug safety and adverse events. Safety assessment is based on cumulative prednisone exposure, the incidence and degree of hypothalamic-pituitary-adrenal axis suppression, and rates of adverse events.

Statistical methods. Analysis of time-to-treatment-failure endpoints and overall survival rate at day-200 post-transplant includes all randomized patients, based on the Kaplan-Meier method and log-rank test, stratified by source of allograft. For each endpoint, the hazard ratio for treatment is estimated based on a Cox proportional hazards model that includes a term for treatment group. Time-to-treatment-failure is right-censored for patients who discontinue study drug during the first 50 days without meeting the criteria for treatment failure, provided the reason for discontinuation was not related to uncontrolled GVHD or study drug-related toxicity. The cumulative probability of treatment failure by Study Days 10, 30, 50, 60, and 80 is estimated by the complement of the Kaplan-Meier estimator. The Z-test is used to compare the rates of treatment failure between groups at each of these time points. Sensitivity analyses are performed using the cumulative incidence method to assess the impact of competing risks. The overall survival rate at day-200 days post-transplant is analyzed in the same manner as described for the treatment failure rates. Because of the variable length of time among patients between transplant and randomization, treatment is defined in the proportional hazards model as a time-dependent covariate. A counting process approach is used to construct the risk set for this analysis. Multivariate models are used to determine if the risk reduction attributed to BDP in the univariate model was still present after accounting for subject-, disease-, and transplant-related factors thought to modify patients' risk of mortality during the 200-day period after transplant. Hypothesis tests of the primary and secondary endpoints are performed using a two-sided significance level of 0.05. No adjustments are made to the significance level for inferential tests of the secondary endpoints. All patients who receive at least one dose of BDP or placebo are included in the assessment of safety. Analyses are done using SAS® (version 8.2) and R (version 2.0.1) software.

ELIGIBILITY:
Inclusion Criteria:

* Allogeneic hematopoietic cell transplant ≥10 days prior to screening
* Symptoms consistent with Grade II intestinal GVHD
* Diagnosis of GVHD confirmed by biopsy
* Confirmed absence of intestinal infection
* Demonstrated ability to swallow 2 tablets of the size and configuration of study drug
* Anti-candidal prophylaxis of the oropharynx
* If female and of childbearing potential, willing to use contraception
* Ability to read, understand, and sign informed consent

Exclusion Criteria:

* Skin GVHD other than a slowly evolving skin rash that involves ≤50% of body surface
* Liver GVHD with total serum bilirubin >3 mg/dL
* Negative intestinal biopsy for GVHD
* Systemic prescription corticosteroid use within 30 days
* Persistent vomiting of oral intake the precludes ingestion of study drug tablets
* Multiorgan failure
* Infection of the mouth or esophagus with a fungal organism
* Known HIV seropositivity
* Pregnancy or lactation
* Previous use of BDP tablets, capsules, or inhalation products
* Use of any investigational drug, biologic, or device within 30 days
* Inability to comply with study procedures and scheduled study visits

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 130
Dates: Start 2001-07; Study Completion 2004-12

PRIMARY OUTCOMES:
Treatment failure (that is, flares of GVHD requiring immunosuppressive drug therapy) at study day 50.

SECONDARY OUTCOMES:
Treatment failure at study day 80.
Survival at transplant day 200.
Adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy C. Rodell, M.D., Study Director — Enteron Pharmaceuticals, Inc., a subsidiary of DOR BioPharma; Scott Cruickshank, Ph.D., Study Director — Enteron Pharmaceuticals Inc, a subsidiary of DOR BioPharma
Locations (1):
- Fred Hutchinson Cancer Research Center, Seattle, Washington, United States

REFERENCES:
- [Background] McDonald GB, Bouvier M, Hockenbery DM, Stern JM, Gooley T, Farrand A, Murakami C, Levine DS. Oral beclomethasone dipropionate for treatment of intestinal graft-versus-host disease: a randomized, controlled trial. Gastroenterology. 1998 Jul;115(1):28-35. doi: 10.1016/s0016-5085(98)70361-0. PMID 9649455
- [Background] Baehr PH, Levine DS, Bouvier ME, Hockenbery DM, Gooley TA, Stern JG, Martin PJ, McDonald GB. Oral beclomethasone dipropionate for treatment of human intestinal graft-versus-host disease. Transplantation. 1995 Dec 15;60(11):1231-8. PMID 8525516
- [Result] Hockenbery DM, Cruickshank S, Rodell TC, McDonald GB. A phase 3 randomized, placebo-controlled study of oral beclomethasone 17, 21-dipropionate (BDP) in conjunction with ten days of high-dose prednisone therapy for patients with gastrointestinal graft vs. host disease. Proceedings of the American Association for Cancer Research 45 (Supplement): 109, 2005. Presented at the annual meeting of the American Association for Cancer Research, Anaheim, CA, 2005.